CLINICAL TRIAL: NCT00962169
Title: Development and Pilot Testing of an Implementation Strategy to Increase Physiotherapists'Adherence to Evidence-based Guideline for Patients With Low Back Pain: a Planned, Systematic and Theory-based Approach
Brief Title: Guideline Implementation in Physiotherapy
Acronym: GIPhT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Radboud University Medical Center (Other)
Collaborators: Maastricht University Medical Center (Other); ZonMw: The Netherlands Organisation for Health Research and Development (Other); The University of Texas Health Science Center, Houston (Other); Royal Dutch Society for Physiotherapy (Unknown); Dutch Institute for Allied Health Care (Unknown)
Responsible Party: Prof. Dr. RAB Oostendorp, University Medical Center St Radboud Nijmegen
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: ZonMw 80-007028-98-07309; CMO 2007/172
Record Dates: First submitted 2009-08-17; First posted 2009-08-19 (Estimated); Last update posted 2009-08-19 (Estimated); Status verified 2009-08

CONDITIONS: Low Back Pain
Keywords: Guideline adherence; Implementation; Physical therapy; Low back pain; Health plan implementation
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Quality improvement program (Experimental)
  Interventions: Other: Behavioral and managerial
- Electronic patient device (EPD) (Experimental)
  Interventions: Other: Behavioral and IT

INTERVENTIONS:
Other: Behavioral and managerial — The quality improvement program is a multi-level intervention program to increase adherence to the Dutch physical therapy Guidelines for Low Back Pain. It consists of two program parts, one for practice quality managers and the other for individual therapists. The management part aims to increase commitment amongst practice owners towards high quality of care, including the appropriate use of guidelines, and addresses the structure and the culture of the physical therapy practice. This part of the program is based on the INK management model and the colour model of De Caluwé. The individual part of the intervention is aimed at increasing physical therapists' guideline adherence by raising awareness and improving recording and clinical reasoning. This part of the intervention is based on psychosocial and educational theories and especially on the principles of Self Regulation.
  Arms: Quality improvement program
Other: Behavioral and IT — The interventions makes use of an improved EPD for physical therapists. Compared to the existing EPDs, the EPD for the present study presents decision information for physical therapists. This decision information is directly based on the recently revised physical therapy guidelines for Low Back Pain and attached to the subsequent steps of clinical reasoning that are inherent to the diagnostic and treatment stages of the usual process of physical therapy care.
  Other Names: FysioDesk EPD.
  Arms: Electronic patient device (EPD)

SUMMARY:
The purpose of this study is 1) to develop an intervention strategy to increase physiotherapists' adherence to evidence-based practice guidelines, 2) to try out this intervention on a small scale to determine what efficacy may be expected from it, and 3) to determine the value of a planned, systematic and theory-based approach that was followed in developing and implementing the intervention.

DETAILED DESCRIPTION:
Summary

The main objective is the planned, systematic, and theory-based development and pilot testing of an intervention strategy to increase physiotherapists' adherence to evidence-based practice guidelines for low back pain. Although it has been demonstrated that the recommendations of these guidelines are effective, its implementation in physiotherapy practice remains limited. This incomplete implementation results in a considerable inefficiency in physiotherapy practice (e.g. the regular use of less effective treatment strategies) and consequently contributes to the extensive socio-economic problems associated with low back pain (1.7% of the BNP). Until now, however, implementation strategies to increase guideline adherence have not been very effective. The lack of a coherent theoretical framework has been pointed out as a possibly important explanatory factor. Recent reports therefore emphasize an expansion of the theoretical basis with regards implementation problems.

The present project (January 2007) will build on the promising results of a cross-sectional study among Dutch physiotherapists, which applied the Precede-Proceed planning model to assess determinants of guideline adherence. To that end, a theoretical framework was constructed that combined the Diffusion of Innovations Theory, the Precaution Adoption Process Model, and elements of Organization Development. The questionnaire based on this framework turned out to be a very useful tool for systematically studying barriers and facilitators associated with guideline adherence. However, a similar, but longitudinal study is needed to assess determinants that actually predict guideline adherence. For this longitudinal study, the framework needs to be slightly revised (5 months). The adapted theoretical framework in turn, will guide the subsequent revision of the determinant questionnaire (3 months).

The longitudinal determinant study (10 months) among primary care physiotherapists (N = 1,600) will be performed via mail. Determinants of guideline adherence will be assessed with the revised questionnaire. Actual guideline adherence will be determined with recently developed longitudinal paper&pencil vignettes that cover the eleven most important indicators of adherence. Statistical analyses of these combined data will disclose which individual, social and / or organizational determinants in fact predict guideline adherence.

The results of the longitudinal study will be used to systematically develop an implementation enhancing strategy (8 months), specifically aimed at modifying the determinants predicting adherence. The development will be based on the Intervention Mapping approach. This approach will, for instance, assists in choosing objectives and strategies of change, and in combining these into a coherent program plan. To assess the efficacy of this combination of implementation strategies, a pilot test (4 months) will be performed among primary care physiotherapists (N = 30) within a network of physiotherapy practices (N = 10). The short-term effects on determinants predicting guideline adherence and on actual guideline implementation will be assessed in a similar way as during the preceding longitudinal study. Additional process information will be collected to refine the implementation enhancing strategy and to explore opportunities for further implementation of this strategy in primary care. A secondary objective of the present study is to further examine the value of the planned, systematic, and theory-based approach for the implementation of practice guidelines in general. Depending on the findings of the present study, we expect to be able to formulate implications for the use of a coherent theoretical framework in the current practice of guideline implementation and in the development of strategies to increase guideline adherence among a wider variety of health care professions, as well as the use of planning models and systematic intervention development models in future implementation efforts and guideline adherence studies.

This study will be the first in the field of guideline implementation that applies (1) a comprehensive theoretical framework for guideline adherence, (2) the Precede-Proceed planning model for the assessment of determinants predicting guideline adherence, and (3) the systematic approach of Intervention Mapping for the development of an implementation strategy. The results will be reported in peer-reviewed articles and included in a dissertation (December 2009).

ELIGIBILITY:
Inclusion Criteria:

Arm 1 Quality improvement program

* Physiotherapy practices that have started or finalized a quality registration procedure (HNK)

Arm 2 Electronic patient device

* Physiotherapists that are acquainted with the use of EPDs in their practice

Exclusion Criteria:

* Physiotherapists enrolled in other quality improvement programs

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2009-07; Primary Completion 2009-12 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
Guideline adherence | 3 months

SECONDARY OUTCOMES:
Determinants of guideline adherence | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Rob Oostendorp, Professor, Study Director — University Medical Center St Radboud Nijmegen
Locations (1):
- IQ healthcare / Radboud UMCN, Nijmegen, Netherlands

REFERENCES:
- [Background] Bekkering GE. Physiotherapy guidelines for low back pain. Development, implementation, and evaluation. Vrije Universiteit Amsterdam, 2004. Fritz JM, Cleland JA, Brennan GP. Does adherence to the guideline recommendation for active treatments improve the quality of care for patients with acute low back pain delivered by physical therapists? Med Care 2007;45(10):973-80. Grimshaw JM, Thomas RE, MacLennan G, Fraser C, Ramsay CR, Vale L, et al. Effectiveness and efficiency of guideline dissemination and implementation strategies. Health Technol Assess 2004;8(6 iii-iv):1-72. Harting J, Rutten GM, Rutten ST, Kremers SP. A Qualitative Application of the Diffusion of Innovations Theory to Examine Determinants of Guideline Adherence Among Physical Therapists. Phys Ther 2009. Rutten G, Kremers S, Rutten S, Harting J. A theory-based cross-sectional survey demonstrated the important role of awareness in guideline implementation. J Clin Epidemiol 2009;62(2):167-176 e1. Rutten GMJ, Harting J, Rutten STJ, Bekkering GE, Kremers SPJ. Measuring physiotherapists' guideline adherence by means of clinical vignettes: a validation study. J Eval Clin Pract 2006;12(5):491-500.